CLINICAL TRIAL: NCT01435473
Title: Clinical Assessment of Thrombosis in Children After Heart Surgery: The CATCH Study
Brief Title: Clinical Assessment of Thrombosis in Children After Heart Surgery
Acronym: CATCH
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Other Study IDs: 1000020203
Record Dates: First submitted 2011-09-08; First posted 2011-09-16 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Thrombosis
Keywords: pediatrics; thrombosis; thromboembolic complications; pediatric cardiac surgery
MeSH Terms: conditions — Thrombosis | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children undergoing heart surgery: The study will follow children undergoing cardiac surgery at The Hospital for Sick Children from pre-consultation, throughout surgery, recovery and post-operative follow-up
  Interventions: Procedure: Cardiac Surgery

INTERVENTIONS:
Procedure: Cardiac Surgery

SUMMARY:
Thromboembolic complications (TCs) are important causes of morbidity and mortality after pediatric cardiac surgery, resulting in longer hospital stay, increased risk of early and late post-surgical complications, early reoperation, neurologic and organ damage, and potentially death. The true incidence of blood clots in pediatric surgical patients is unknown.

The overarching objective of this study is to further our understanding of TCs, including quantification, characterization and risk stratification. This study will ultimately allow the development of effective tools for prevention and early identification of TCs, rather than focusing on treatment alone.

DETAILED DESCRIPTION:
There is very limited data on TCs associated with cardiac surgery in pediatric patients. The actual incidence of TCs in this context is not currently known reflecting a lack of clinical suspicion, reporting biases, and/or the use of inappropriate diagnostic tests

Pediatric cardiac surgery is associated with disruption of blood flow, platelet dysfunction and activation, and blood hypercoagulability; all of which are contributing to clot formation

All congenital heart defects are associated with blood flow disturbance but some are associated with more extreme disturbances. The investigators hypothesize that not all types of CHD repairs will be at the same risk of TCs based on the extent of blood flow disturbances they cause. The investigators hypothesize that line location, difficulties in line insertion, including multiple insertion attempts and longer duration of indwelling will be associated with increased risk of TCs.

Pediatric cardiac surgery is associated with inflammation and platelet activation, both of which are potent contributors to blood hypercoagulability: CPB presents a hemostatic challenge associated with an abundance of pro-thrombotic risk factors and an opposite presence of pro-hemorrhagic risk factors. The investigators hypothesize that factors associated with increased platelet activation and inflammation, and in consequence, greater laboratory values of markers of platelet activation and inflammation, will be associated with increased risk of TCs.

Coagulation system activity in children is immature, hyporeactive and exhibits a high degree of resistance to heparin and anticoagulation. The investigators theorize that lower levels of coagulation system activity, presence of high-risk genetic polymorphisms, greater CPB hemodilution, increased heparin requirement and lower blood heparin activity expressed by anti-factor X activity (anti-Xa) concentration during CPB and greater requirement for allogeneic blood will be associated for increased risk of TCs.

There is a lack of consensus on clinical and laboratory signs/symptoms of active thrombosis and on which patients should be routinely screened for TCs. One of the most difficult aspects in the management of TCs is the fact that many episodes are asymptomatic or have non-specific symptoms. Creating a risk stratification model including both clinical and laboratory abnormalities which could be indicative of TCs in the post-operative period in order to identify patients who should undergo more targeted screening is the third aim of this study.

Many methods of TC management have limited effectiveness while highly effective methods are often associated with much risk. The use of thrombolytics in children is rare and only partially effective in many cases. The margin of safety for treatment is thought to be very narrow; the reported frequency of major bleeding episodes varies from 5% to 40%.

Outcomes of TCs are suboptimal, early surgical and long-term complications for survivors are frequent. The creation of risk stratification models for suboptimal surgical outcomes, PTS syndrome and, lower functional health status after surgery will be the fourth and final aim of this study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for cardiac surgery requiring cardiopulmonary Bypass

Exclusion Criteria:

* Known severe risk factors to thromboembolic complications
* Active cancer
* Congenital coagulopathy (e.g. haemophilia)
* No planned cardiology follow-up at the Hospital for Sick Children

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children Undergoing Pediatric Heart Surgery at the Hospital for Sick Children who agree to participate in the CATCH research study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Thromboembolic Complications (TC) after pediatric cardiac surgery | Outcome will be recorded throughout the duration of the participants hospital stay, an expected average of 10 days
  Thrombosis will be recorded through review of post-operative clinical assessments, targeted laboratory testing for blood abnormalities and echocardiographic/ultrasound evaluation.

SECONDARY OUTCOMES:
Assessment of the patients' coagulation, hemostatic and inflammatory system activity | Baseline
  Standard coagulation panel to assess the function of the coagulation system in order to identify the degree of maturity, potential for resistance to anticoagulation and overall activity of the coagulation system.
Genome-Wide Association Study (GWAS) | Baseline
  To identify genetic polymorphisms associated with coagulation system activity, sensitivity and overall thrombotic risk.
Post-operative sign and symptoms of thrombosis | Up to 10 days after surgery
  Daily clinical assessment of signs and symptoms of thrombosis
Post-thrombotic Syndrome (PTS) Evaluation | Up to 2 years after surgery
  Assessment of upper and lower limbs based on the adaptation of the Khule scale. PTS will be classified as mild, moderate and severe.
Neurodevelopment and functional health assessment | Up to 2 years post- surgery
  Subject will undergo Ages and Stages (ASQ, Child Health Questionnaires and PedsQL)
Response of the patients coagulation, hemostatic and inflammatory system activity to cardiopulmonary bypass | Up to 10 days after surgery
  Repeat of complete blood count, inflammatory markers, coagulation and fibrolnolytic systems activity
Proportion of patients with thrombo-occlusive complications of thrombosis | 18-24 months after surgery
  Following events associated with thrombosis:
  * Death / cardiorespiratory arrest associated with thrombosis
  * Embolism (cardioembolic stroke, pulmonary embolism)
  * Obstruction (sinovenous stroke, SVC syndrome)
  * Unanticipated procedures directed at thrombosis or its clinical impact
  * Escalation of antithrombotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Brian W McCrindle, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada